CLINICAL TRIAL: NCT05142176
Title: Bilateral Erector Spinae Plane Block for Management of Acute Postoperative Pain After Pediatric Cardiac Surgeries Through a Midline Sternotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Mogahed, Associate professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 34774/7/21
Record Dates: First submitted 2021-11-06; First posted 2021-12-02 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-12

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Intervention Model Description: Bilateral erector spinae block
Who Masked: Participant, Care Provider
Masking Description: Patients unaware and care giver were unaware about what is injected inthe catheters
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): will receive general anesthesia with bilateral sham erector spinae plane block at the level of T6 transverse process using 0.3 ml/kg normal saline on each side.
  Interventions: Other: Erector spinae catheters insertion; Drug: Postoperative pain management
- Erector spinae plane block group (Active Comparator): will receive bilateral ultrasound-guided erector spinae plane block at the level of T6 transverse process using 0.3 ml/kg bupivacaine 0.25% (on each side) with a maximum dose of 2 mg/kg.
  Interventions: Other: Erector spinae catheters insertion; Drug: Postoperative pain management

INTERVENTIONS:
Other: Erector spinae catheters insertion — Ultrasound-Guided ESPB The ESPB will be performed with the child in a right lateral decubitus position under aseptic precautions by a high frequency (6-13 MHz) linear ultrasound transducer
Drug: Postoperative pain management — IV acetaminophen 15 mg/kg every 8 hours as a component of multimodal analgesia.

SUMMARY:
Many analgesic modalities have been investigated in pediatrics. The analgesic efficacy of bilateral ultrasound-guided erector spinae plane block in pediatric patients undergoing open midline sternotomy will be examined. Methods: 60 patients aged 3- 12 years will be randomly assigned into two groups: Control group will receive general anesthesia with bilateral sham erector spinae plane block at the level of T6 transverse process using 0.3 ml/kg normal saline on each side. Erector spinae plane block group will receive bilateral ultrasound-guided erector spinae plane block at the level of T6 transverse process using 0.3 ml/kg bupivacaine 0.25% (on each side) with a maximum dose of 2 mg/kg. The postoperative pain was assessed using Modified Objective Pain Scores (MOPS) which will be evaluated at 0, 1, 2, 4, 6, 8, 10, and 12 hours after extubation, total consumption of intraoperative fentanyl (1µg/kg IV in case of inadequate analgesia), time to first rescue analgesic administration and postoperative paracetamol consumption will be recorded over the first 24 hours postoperatively.

DETAILED DESCRIPTION:
75 children with an American Society of Anesthesiologists physical status class I and II undergoing cardiac surgical procedures through midline sternotomy . The patients with preoperative ejection fraction <35%, low-cardiac-output syndrome, recurrent ventricular arrhythmias, preoperative inotropic support, allergic to the amide type of local anesthetics (LA), requiring intubation for more than 3 hours or re-exploration, and requiring redo or emergency surgery will be excluded from the study. The enrolled children will be subsequently randomized into 2 groups using a computer generated random number table: Control group will receive general anesthesia with bilateral sham erector spinae plane block at the level of T6 transverse process using 0.3 ml/kg normal saline on each side. Erector spinae plane block group will receive bilateral ultrasound-guided erector spinae plane block at the level of T6 transverse process using 0.3 ml/kg bupivacaine 0.25% (on each side) with a maximum dose of 2 mg/kg. The postoperative pain will be managed with rescue intravenous (IV) fentanyl. Both the groups will receive IV acetaminophen 15 mg/kg every 8 hours as a component of multimodal analgesia. A routine preoperative assessment will be performed for all the patients. Premedication in the form of 1 mg/kg promethazine syrup will be administered, 1 hour before shifting to the operating room. Standard American Society of Anesthesiologists monitoring will be instituted and the children were anesthetized as per institutional protocol. The protocol constituted an induction with sevoflurane in oxygen 50% and air, peripheral IV cannulation of appropriate size followed by IV midazolam, 0.05 to 0.1 mg/kg, fentanyl, l to 2 mg/kg, and rocuronium, 0.6 mg/kg, to facilitate endotracheal intubation. Femoral arterial access will be established for intra-arterial pressure monitoring. Central venous catheter will be inserted in the right internal jugular vein for central venous pressure monitoring in addition to the temperature, end-tidal carbon dioxide, and near infrared spectroscopy monitoring. Anesthesia will be maintained with sevoflurane (0.9-2%) in 50% oxygen in air mixture and supplemental boluses of 0.1 mg/kg of atracurium, with the hemodynamics maintained within 20% of the baseline. Ultrasound-Guided ESPB The ESPB will be performed with the child in a right lateral decubitus position under aseptic precautions. A high frequency (6-13 MHz) linear ultrasound transducer (Sonosite Inc, Bothell WA) was placed in a longitudinal orientation over the T3 transverse process lateral to the spinous process. After identifying the muscles (trapezius, rhomboid major, and erector spinae) above the hyperechoic transverse process image, a 5-cm 22- guage Stimuplex A block needle (B. Braun, Melsungen, Germany) will be inserted in-plane in a cephalo-caudad direction. The endpoint will be defined as the needle pointing to the tip of transverse process piercing the erector spinae muscle. The LA will be deposited at this position, close to the costotransverse foramen. The needle tip position will be confirmed by hydrolocation with 0.5 to 1 mL of 1% lidocaine indicating linear fluid spread lifting the fascial plane between the transverse process and erector spinae muscle. After careful negative aspiration, 1.5 mg/kg of 0.2% ropivacaine will be administered under ultrasound guidance . The process will be repeated with injection of 0.3 ml/kg bupivacaine 0.25%bupivacaine on the contralateral side adding up to a cumulative dose of 2 mg/kg ropivacaine. Following sternotomy, adequate heparinization will be achieved with a resultant activated clotting time >480 seconds before the initiation of cardiopulmonary bypass in both the groups. After a satisfactory surgical correction, the patient will be weaned off cardiopulmonary bypass followed by protamine administration. The patients will be transferred to the intensive care unit (ICU) after completion of the procedure.

Postoperative ICU Management and Postoperative Pain Assessment The electrocardiogram, invasive blood pressure, respiratory rate, and pulse oximetry (Spo2) were monitored and recorded throughout the postoperative period. The study subjects will be extubated within 2 to 3 hours postoperatively once the exubation criteria (conscious, hemodynamically stable, (peak inspiratory pressure) PIP <20 cmH2O above positive end-expiratory pressure (PEEP)will be fulfilled, no neuromuscular blockade, and normal arterial blood gas analysis). Postoperative pain assessment will be performed using Modified Objective Pain Score (MOPS)9 at 0, 1, 2, 4, 6, 8, 10, and12hours post extubation. Acetaminophen, 15 mg/kg, IV, every 8 hours will be administered in both the groups. . A rescue analgesic fentanyl, 0.5 to 1 mg/kg, will be administered when the MOPS score was≥ 4 at rest. Postoperative adverse effects such as nausea, vomiting, cardiac arrhythmia, and complications such as LA toxicity, and vascular puncture were recorded and treated. Statistical Analysis Primary and Secondary Endpoints MOPS at 0, 1, 2, 4, 6, 8, 10, and 12 hours post extubation constituted the primary endpoints. The secondary endpoints will include intraoperative fentanyl requirement, extubation time, time to first rescue analgesic requirement, postoperative cumulative fentanyl requirement up to 12 hours, Ramsay sedation score, ICU stay, and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* children undergoing cardiac surgical procedures through midline sternotomy

Exclusion Criteria:

* The patients with preoperative ejection fraction <35%
* allergic to the amide type of local anesthetics (LA)
* preoperative inotropic support

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2022-02-05 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Modified Objective Pain Score (MOPS)0 | at immediately post extubation.
  A rescue analgesic fentanyl, 0.5 to 1 mg/kg, will be administered when the MOPS score was≥ 4 at rest
Modified Objective Pain Score (MOPS)1 | at1 hour post extubation.
  A rescue analgesic fentanyl, 0.5 to 1 mg/kg, will be administered when the MOPS score was≥ 4 at rest
Modified Objective Pain Score (MOPS)2 | at 2 hour post extubation.
  A rescue analgesic fentanyl, 0.5 to 1 mg/kg, will be administered when the MOPS score was≥ 4 at rest
Modified Objective Pain Score (MOPS)3 | at 4 hour post extubation.
  A rescue analgesic fentanyl, 0.5 to 1 mg/kg, will be administered when the MOPS score was≥ 4 at rest
Modified Objective Pain Score (MOPS)4 | at 6 hour post extubation.
  A rescue analgesic fentanyl, 0.5 to 1 mg/kg, will be administered when the MOPS score was≥ 4 at rest
Modified Objective Pain Score (MOPS)5 | at 8 hour post extubation.
  A rescue analgesic fentanyl, 0.5 to 1 mg/kg, will be administered when the MOPS score was≥ 4 at rest
Modified Objective Pain Score (MOPS)6 | at 12 hour post extubation.
  A rescue analgesic fentanyl, 0.5 to 1 mg/kg, will be administered when the MOPS score was≥ 4 at rest